CLINICAL TRIAL: NCT03094806
Title: Vibratory/Positive Expiratory Pressure Device and Hospital Length of Stay for Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Vibratory PEP Device and Hospital Length of Stay for Acute Exacerbation of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Jeremy Weingarten, MD, Dr, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 470455
Record Dates: First submitted 2015-05-27; First posted 2017-03-29 (Actual); Results first posted 2018-10-11 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acapella Vibratory PEP Therapy Device (Experimental): Subject will use the device 3 times a day throughout hospital stay
  Interventions: Device: Acapella Vibratory PEP Therapy Device plus usual care
- Sham Acapella Vibratory PEP Device (Placebo Comparator): Subject will use the sham device 3 times a day throughout hospital stay
  Interventions: Device: Sham Acapella Vibratory PEP Device plus usual care

INTERVENTIONS:
Device: Acapella Vibratory PEP Therapy Device plus usual care — The acapella® Vibratory PEP Therapy System (PEP-FV) device is a handheld device that operates in same principle as standard FV. Unlike standard FV, it is not gravity dependent. It comes in two different devices to accommodate for different flows rates of the patient. It has similar properties of a standard FV and may be better tolerated.
  Arms: Acapella Vibratory PEP Therapy Device
Device: Sham Acapella Vibratory PEP Device plus usual care — The Sham Acapella Vibratory PEP Device is the same as the Therapy Device, except the flutter valve has been removed from the device.
  Arms: Sham Acapella Vibratory PEP Device

SUMMARY:
This study is evaluating the use of a respiratory device, the Acapella Vibratory Positive Expiratory Pressure (PEP) Therapy device, in patients admitted to the hospital with a chronic obstructive pulmonary disease (COPD) exacerbation.

DETAILED DESCRIPTION:
The investigators hypothesize that the PEP-FV used as adjunctive therapy in patients hospitalized for an acute exacerbation of COPD will result in decreased hospital length of stay and improvement of overall COPD-related health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with COPD exacerbation as a primary diagnosis
* Subjectively produces more than 1 tablespoon (15 ml) / day of sputum
* Has the subjective feeling that he/she cannot cough up or clear her secretions
* Physical respiratory system exam by the physician with evidence of course ronchi suggestive of impacted secretions
* > 10 pack-year smoking history

Exclusion Criteria:

* Cannot use the flutter device or unable to follow commands
* Altered mental status
* Known active malignancy
* Known systolic congestive heart failure (CHF) with ejection fraction (EF) < 40% or clinically in acute CHF exacerbation as documented by cardiologist or primary diagnosis other than COPD
* Pregnancy
* Patients in severe exacerbation (Intubated, Continuous use of NIPPV, Unable to speak full sentences)
* Intracranial pressure (ICP) >20 mmHg
* Hemodynamic instability (requiring vasopressor support)
* Recent facial, oral, or skull surgery or trauma.
* Acute sinusitis.
* Epistaxis.
* Esophageal surgery.
* Active Hemoptysis (More than 2 tablespoons of frank blood per day)
* Nausea.
* Severe earache or discharge from ear. (Known or suspected tympanic membrane rupture or other middle ear pathology)
* Untreated pneumothorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Weingarten, MD, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

REFERENCES:
- [Derived] Milan S, Bondalapati P, Megally M, Patel E, Vaghasia P, Gross L, Bachman EM, Chadha P, Weingarten JA. Positive Expiratory Pressure Therapy With And Without Oscillation And Hospital Length Of Stay For Acute Exacerbation Of Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2019 Nov 20;14:2553-2561. doi: 10.2147/COPD.S213546. eCollection 2019. PMID 31819393

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Started | 44 | 47
Completed | 44 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device | Total
Number analyzed (Participants) | 44 | 47 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 20 | 48
  >=65 years | 16 | 27 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.6) | 65.9 (12.2) | 64.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 15 | 18 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 18 | 31
  White | 31 | 29 | 60
  More than one race | NA — not measured | NA — not measured | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — not measured | NA — not measured | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 44 | 47 | 91
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.6 (11.9) | 30.7 (8.2) | 32.6 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: Time of admission to time of discharge from hospital
Time Frame: Up to 2 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Number analyzed (Participants) | 44 | 47
days | 4.8 [3.9 to 6.1] | 3.2 [3.0 to 4.3]

2. Secondary Outcome: Analysis of Change in Daily Sputum Production
Description: Sputum production in a 24 hour period in mL volume
Time Frame: Up to 5 days
Measure: Mean (Standard Deviation); unit: volume in mL
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Number analyzed (Participants) | 44 | 47
volume in mL
  Sputum production day 1 | 6.6 (8.8) | 14.6 (17.6)
  Sputum production day 2 | 7.5 (8.5) | 15.9 (16.8)
  Sputum production day 3 | 6.5 (6.7) | 15.9 (16.6)
  Sputum production day 4 | 5.3 (7.0) | 13.4 (16.4)
  Sputum production day 5 | 2.9 (5.7) | 13.3 (15.9)

3. Secondary Outcome: Dyspnea on the Borg Scale
Description: Scale is used to rate the difficulty of breathing. It starts at 0 where the breathing is causing no difficulty at all and progresses through to number 10 where the breathing difficulty is maximal.
Time Frame: Up to 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Number analyzed (Participants) | 44 | 47
score on a scale
  Borg scale day 1 | 5.0 (2.4) | 5.1 (2.5)
  Borg scale day 2 | 3.7 (2.1) | 4.3 (2.5)
  Borg scale day 3 | 3.3 (2.2) | 3.3 (2.2)
  Borg scale day 4 | 2.9 (2.1) | 3.3 (2.5)
  Borg scale day 5 | 3.1 (2.4) | 3.2 (2.0)

4. Secondary Outcome: Dyspnea on the MMRC Scale
Description: The Modified Medical Research Council (MMRC) dyspnea scale is used to assess an individual's shortness of breath. It starts at 0 where the shortness of breath occurs during strenuous exercise and progresses through to number 4 where the shortness of breath is maximal.
Time Frame: Up to 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Number analyzed (Participants) | 44 | 47
score on a scale
  MMRC scale day 1 | 2.2 (1.0) | 2.4 (1.3)
  MMRC scale day 2 | 1.9 (1.0) | 2.1 (1.4)
  MMRC scale day 3 | 1.7 (1.0) | 2.2 (1.4)
  MMRC scale day 4 | 1.7 (1.0) | 2.2 (1.3)
  MMRC scale day 5 | 1.8 (1.0) | 2.4 (0.9)

5. Secondary Outcome: Change in 6MWT Test
Description: A six-minute walk test (6MWT) measures the distance that an individual can walk on a flat, hard surface in a period of six minutes. This is used to assess the exercise tolerance measured by the difference in meters between the tests.
Time Frame: Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Number analyzed (Participants) | 44 | 47
meters
  6MWT day 1 | 168.8 (118.9) | 206.7 (120.8)
  6 MWT day 5 | 200.1 (90.3) | 199.3 (119.9)

6. Secondary Outcome: Difference in Bedside Spirometry
Description: Degree of airflow obstruction (FEV1/FVC)
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Number analyzed (Participants) | 44 | 47
ratio | 70.7 (20.6) | 57.7 (13.8)

7. Secondary Outcome: In Hospital Mortality
Description: Death at the time of discharge
Time Frame: Up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Number analyzed (Participants) | 44 | 47
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Admission to discharge or Day 5, whichever occurred first.
Arm/Group | Acapella Vibratory PEP Therapy Device | Sham Acapella Vibratory PEP Device
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/47
Other Adverse Events (participants affected / at risk) | 0/44 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No